CLINICAL TRIAL: NCT07140367
Title: "Transarterial Microembolization (TAME) in Inflammatory Knee Pathology: Prospective Observational Study."
Brief Title: "Transarterial Microembolization (TAME) in Inflammatory Knee Pathology"
Acronym: TAME-OA
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Giancarlo Facchini, MD PhD, Istituto Ortopedico Rizzoli
Other Study IDs: CE AVEC: 350/2025/Oss/IOR
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Articular Diseases; Knee Osteoarthristis
Keywords: embolization; transarterial microembolization; TAME; arthritis; inflammatory articular disease; arthropathy; knee; osteoarthritis
MeSH Terms: conditions — Arthritis; Joint Diseases; Osteoarthritis | interventions — Embolization, Therapeutic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Performed microembolization
  Interventions: Procedure: Transarterial Microembolization

INTERVENTIONS:
Procedure: Transarterial Microembolization — Identification of the hypervascularization of the knee. Selective and super-selective catheterization of pathological genicular arterial branches, through the use of micro-catheters. - Injection of embolizing material (Nexsphere-F - Kardia) - Control of technical success: the embolization will be followed by diagnostic arteriography that will evaluate the success of the procedure (occlusion of more than 90 percent of the pathologic vasculature).
  Other Names: TAME; embolization; transarterial embolization

SUMMARY:
Patients with knee OA and chronic pain refractory to at least 3 months of conventional conservative therapy will be included in the study, which will evaluate the clinical results obtained after treatment with selective arterial embolization (selection and enrollment, treatment with selective arterial embolization, follow-up checks). Forty-three patients will be included in the study and will undergo the transarterial microembolization procedure after signing the informed consent form for participation in the study and the collection of anamnestic data. Subsequently, patients will be followed up with clinical evaluation at 1, 3, 6, 12, and 24 months of follow-up or until possible dropout for other treatment.

DETAILED DESCRIPTION:
Degenerative and inflammatory joint disease is a common and debilitating condition that causes pain and limited mobility, with osteoarthritis (OA) being the most common form. The knee is the most commonly affected joint, with an estimated 600 million people worldwide currently living with unilateral or bilateral knee OA, marking a 113% increase since 1990. Although risk factors include obesity, advanced age, and female gender, most individuals are susceptible to the pathophysiological cascade of OA, which likely explains the dramatic global burden of the disease and its associated economic consequences. These joint disorders have a significant impact on individuals' quality of life. When they occur in mild or moderate form, a series of therapeutic strategies can be implemented, but these rarely lead to a significant reduction in pain and do not alter the course of the disease. Standard treatment includes exercise, postural measures, weight control, and pharmacotherapy. Intra-articular injections of hyaluronic acid or platelet-rich plasma (PRP) have emerged as new non-surgical treatment options. Surgical joint replacement is reserved for the most severe cases, with intense pain and functional disability. However, many patients suffer from refractory chronic pain, are not candidates for surgery, or refuse it. In addition, some patients may experience complications associated with long-term pharmacotherapy, such as renal or hepatic failure, opioid dependence, or local problems resulting from injections, such as infections. In recent years, geniculate artery embolization has emerged as a promising option for patients with knee pain due to OA who are refractory to conservative therapies and who are not eligible for or choose not to undergo arthroplasty surgery.

Patients with knee OA and chronic pain refractory to at least 3 months of conventional conservative therapy will be included in the study, which will evaluate the clinical results obtained after treatment with selective arterial embolization (selection and enrollment, treatment with selective arterial embolization, follow-up checks). Forty-three patients will be included in the study and will undergo the transarterial microembolization procedure after signing the informed consent form for participation in the study and the collection of anamnestic data. Subsequently, patients will be followed up with clinical evaluation at 1, 3, 6, 12, and 24 months of follow-up or until possible dropout for other treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients with degenerative knee disease:

1. Age over 40 years;
2. Moderate knee OA (grade 2-3 according to the Kellgren-Lawrence score) for which an indication for total knee arthroplasty surgery has already been given;
3. Knee OA with an inflammatory component (night pain, pain at rest, recurrent episodes of effusion, swelling and/or redness);
4. Persistent and moderate or severe knee pain (VAS score > 4);
5. Failure after at least 3 months of conservative therapies (e.g., physical therapy, drug therapy with NSAIDs and pain relievers, hyaluronic acid infiltration, corticosteroids, or orthobiologics).
6. Signature of informed consent
7. Case declared eligible for treatment following discussion at internal multidisciplinary meeting on degenerative-inflammatory disease

Exclusion Criteria:

1. Mentally incompetent patients;
2. Patients with trauma in the 6 months prior to treatment;
3. Patients with malignant neoplasms;
4. Patients with rheumatic diseases;
5. Patients on anticoagulant-antiaggregant therapy (including if therapy can be discontinued 5 days earlier);
6. Patients abusing alcoholic beverages, drugs, or medications;
7. Patients undergoing surgery of the affected knee in the previous 12 months;
8. INR <2;
9. Platelet count <30,000;
10. Renal function: GFR<30ml/min;
11. Pregnancy;
12. Allergy to iodinated contrast.
13. Ineligibility to perform MRI examination.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by inflammatory arthropathy of the knee who underwent genicular artery microembolization.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain (VAS score) | 1 year
  Clinical assessment regarding pain by Visual Analogue Scale (VAS) score (0-100 mm), in which 0 represents no pain, and 100 represents maximum pain imaginable.

SECONDARY OUTCOMES:
Improvement in quality of life (SF-36) | 2 years
  Clinical assessment regarding quality of life by SF-36 questionnaire. The SF-36 is a widely used tool to measure health-related quality of life. It has 36 questions covering 8 domains: Physical Functioning, Role Limitations due to Physical Health, Bodily Pain, General Health, Vitality, Social Functioning, Role Limitations due to Emotional Problems, Mental Health.
  Plus, there is one item on health change over the past year.
  Scoring:
  Once items are recoded so that higher scores always = better health, domain scores are computed by averaging item scores, then transforming to a 0-100 scale (0 = worst health, 100 = best).
Pain, stiffness, and physical functioning of the joints (WOMAC score) | 2 years
  It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68), which mainly concern daily activities (e.g., getting up from a sitting position, bending over, going up and down stairs, etc.). The score is then normalized on a scale of 0-100. Higher values indicate a worse outcome.
Range of motion | 2 years
  Objective parameter used to assess joint mobility and functional ability.
  - Good/Normal ROM:
  Extension: 0° (up to -5°/-10° hyperextension can be physiological).
  Flexion: 130°-150°.
  - Clinically acceptable ("good enough" for daily life):
  Flexion >120°.
  Full extension (0°) is essential; even small deficits are significant.
  - Reduced:
  Flexion <110°.
  Extension loss >5°.
Overall assessment of treatment | 2 years
  The patient will be asked to indicate their level of satisfaction (on a scale from 0 to 10) with the treatment received at each follow-up visit during the clinical trial.
Bilateral Trans- and Suprapatellar Circumferences | 2 years
  To compare muscle mass and joint swelling/edema between the injured and non-injured side.
  * Good/Normal: difference ≤1 cm between sides.
  * Borderline/Reduced: difference 1.5-2 cm → may indicate muscle atrophy or swelling.
  * Significant abnormality: >2 cm difference.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
Privacy concerns

REFERENCES:
- [Background] Sapoval M, Querub C, Pereira H, Pellerin O, Boeken T, Di Gaeta A, Ahmar MA, Lefevre-Colau MM, Nguyen C, Daste C, Lacroix M, Laredo JD, Sabatier B, Martelli N, Chatellier G, Dean C, Rannou F. Genicular artery embolization for knee osteoarthritis: Results of the LipioJoint-1 trial. Diagn Interv Imaging. 2024 Apr;105(4):144-150. doi: 10.1016/j.diii.2023.12.003. Epub 2023 Dec 14. PMID 38102013
- [Background] Little MW, O'Grady A, Briggs J, Gibson M, Speirs A, Al-Rekabi A, Yoong P, Ariyanayagam T, Davies N, Tayton E, Tavares S, MacGill S, McLaren C, Harrison R. Genicular Artery embolisation in Patients with Osteoarthritis of the Knee (GENESIS) Using Permanent Microspheres: Long-Term Results. Cardiovasc Intervent Radiol. 2024 Dec;47(12):1750-1762. doi: 10.1007/s00270-024-03752-7. Epub 2024 May 31. PMID 38819473
- [Background] Okuno Y, Korchi AM, Shinjo T, Kato S. Transcatheter arterial embolization as a treatment for medial knee pain in patients with mild to moderate osteoarthritis. Cardiovasc Intervent Radiol. 2015 Apr;38(2):336-43. doi: 10.1007/s00270-014-0944-8. Epub 2014 Jul 4. PMID 24993956